CLINICAL TRIAL: NCT05941689
Title: Research on the Auxiliary Diagnosis and Treatment System of Digestive Endoscopy Based on Artificial Intelligence: An Efficacy Study of Artificial Intelligence-assisted Colonic Polyp Detection System
Brief Title: Efficacy of Artificial Intelligence-assisted Colonic Polyp Detection System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 202306499
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-07

CONDITIONS: Adenoma Colon

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-assisted group (Experimental): Subjects in this group undergo AI-assisted colonoscopy. The AI-assisted system not only has the function of automatic polyp detection, but also has the function of colonoscopy quality control.
  Interventions: Device: AI-assisted colonoscopy
- control group (No Intervention): Subjects in this group undergo routine colonoscopy.

INTERVENTIONS:
Device: AI-assisted colonoscopy — AI can not only detect suspicious lesions timely, and label them in the field of view of the colonoscopy, but also monitor withdrawal speed and calculate the clean withdrawal time automatically.
  Arms: AI-assisted group

SUMMARY:
This is a randomized controlled multicenter clinical trial of computer-aided detection (CADe) system for the adjuvant diagnosis of intestinal polyps/adenomas ever conducted in a Chinese population. In addition, this study will evaluate the effect of CADe system on adenoma detection of endoscopists under fatigue.

ELIGIBILITY:
Inclusion Criteria:Patients who need to undergo colonoscopy. -

Exclusion Criteria:Patients with CRC, inflammatory bowel disease, previous colonic resection, and antithrombotic therapy precluding polyp resection were excluded.

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1906 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
adenoma detection rate | up to 2months
  The proportion of patients with at least one histologically proven adenoma or carcinoma
withdrawal time compliance rate | up to 2months
  The proportion of patients with clean withdrawal time >6min.

SECONDARY OUTCOMES:
polyp detection rate | up to 2 months
  The proportion of patients with at least one polyp.
adenoma per colonoscopy | up to 2 months
  The number of adenomas detected per colonoscopy
polyp per colonoscopy | up to 2 months
  The number of polys detected per colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowei Liu, doctor, Principal Investigator — Xiangya Hospital of Central South University
Locations (2):
- China (2):
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Loudi Central Hospital, Loudi, Hunan